CLINICAL TRIAL: NCT06503861
Title: Southern Indiana Farm to Health Initiative: Evaluation of Produce Prescription Intervention
Brief Title: Community-designed Food Is Medicine for Adults With Diabetes
Acronym: FarmtoHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Julia Valliant, Assistant Research Scientist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002563351; IU-IIR-FARM2HEALTH (Other: IU Office of Clinical Research)
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Is Medicine intervention (Experimental)
  Interventions: Behavioral: Food Is Medicine intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Food Is Medicine intervention — The intervention provides regular meal kits as well as cooking and nutritional education.
  Arms: Food Is Medicine intervention

SUMMARY:
The goal of this clinical trial is to learn if an educational intervention can affect clinical outcomes in adults with diabetes. The main question it aims to answer is:

Can a Food Is Medicine intervention affect obesity and/or diabetes markers in adults?

Researchers will compare a Food Is Medicine arm to a control arm to answer the research question.

Participants will provide biometrics and questionnaire responses at three time points. Those in the Food Is Medicine arm will receive regular free meal kits combined with cooking and nutritional education.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years, weight 100+ pounds, HbA1c >7% in 2020

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
Participants' diabetes level or severity | Three time points over approximately 9 months (time1 baseline, time 2 post-intervention, time 3 long-term)
  Participants' glycated hemoglobin - Hemoglobin A1c (HbA1c)
Participants' obesity level or severity | Three time points over approximately 9 months (time1 baseline, time 2 post-intervention, time 3 long-term)
  Body mass index (BMI)

SECONDARY OUTCOMES:
Dietary behaviors | Three time points over approximately 9 months (time1 baseline, time 2 post-intervention, time 3 long-term)
  Self-reported food consumption frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Julia CD Valliant, PhD, Principal Investigator — Indiana University
Locations (1):
- Southern Indiana Community Health Care, Paoli, Indiana, United States

IPD SHARING:
Plan to Share IPD: No